CLINICAL TRIAL: NCT02487927
Title: The Classification of Difficult Weaning and the Predictive Value of Relative Factors for Difficult Weaning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, Professor, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: Weaning Study
Record Dates: First submitted 2015-06-23; First posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Intensive Care Medicine; Mechanical Ventilation; Weaning
MeSH Terms: interventions — Weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Weaning success: patients pass SBT and weaning without any ventilation in 48 hours
  Interventions: Behavioral: weaning
- weaning failure: patients do not pass SBT or ventilation with any ventilation in 48 hours
  Interventions: Behavioral: weaning

INTERVENTIONS:
Behavioral: weaning — T piece

SUMMARY:
To evaluate the distribution of different types of difficult weaning and the predictive value of weaning relative factors.

DETAILED DESCRIPTION:
108 patients who passed the spontaneous breathing test (SBT) were included in this study,every patient were performed 30-60 minutes SBT after enrollment.Patients were divided into succeed weaning and difficult weaning group according the results of SBT, the difficult weaning group were futher divided into A(Airway and Lung dysfunction),B（Brain dysfunction）,C（Cardic dysfunction）,D（Diaphragm dysfunction）,E（Endocrine and metabolic dysfunction）five different groups according to the causes of difficult weaning. The respiratory mechanical parameters,the diameter of inferior vena cava and the diaphgram excursion were recorded before SBT and 30 minutes after SBT.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation patients
* prepared to weaning
* sign on the acknowledged

Exclusion Criteria:

* endotracheotomy
* single lung
* pregnant
* heart,liver,renal failure

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: mechanical vetilation patients in ICU, and the patients are weaninng candidates
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
the reasons of difficult weaning | 30 mins

SECONDARY OUTCOMES:
The predictive value of diaphragm associated values in weaning | 30mins

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, Dr, Study Director — Southeast University
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China